CLINICAL TRIAL: NCT03537131
Title: Dapagliflozin During Exercise for the Prevention of Hypoglycaemia in Type 1 Diabetes
Brief Title: Dapagliflozin During Exercise for the PrevenTion of Hypoglycaemia
Acronym: DEPTH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Temporary halt due to COVID-19 pandemic
Sponsor: University of Oxford (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Oxford Brookes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23092017; 2017-003911-21 (EudraCT Number)
Record Dates: First submitted 2018-04-25; First posted 2018-05-25 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; dapagliflozin; exercise; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Motor Activity; Hypoglycemia | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm B1- Dapagliflozin once only dose (Active Comparator): Participants who will take one tablet of Dapagliflozin 10 mg on the day of the exercise challenge.
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet
- arm B2- Dapagliflozin daily administration (Active Comparator): Participants who will take a daily dose of Dapagliflozin 10 mg before and after the exercise challenge.
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet — taken once a day
  Other Names: forxiga

SUMMARY:
There are approximately 400,000 people in the UK who are living with type 1 diabetes (T1DM), of whom 29,000 are children.

People with T1DM experience on average 2 episodes of symptomatic hypoglycaemia per week , and exercise (especially aerobic) increases this risk . Strategies to prevent hypoglycaemia during and after exercise include increasing glucose consumption and reducing insulin dose, however overcompensation may result in worsening of blood glucose control.

Dysregulated glucagon secretion, manifested as a reduced counter-regulatory response during hypoglycaemia, is a key feature in T1DM, occurring soon after diagnosis.

Anecdotal evidence suggests that SGLT-2 (sodium/glucose cotransporter-2) inhibitors (SGLT2i) such as dapagliflozin prevent exercise-induced hypoglycaemia in T1DM. SGLT2is promote glucose excretion without causing hypoglycaemia.Paradoxically, given their mode of action, they increase plasma glucose and stimulate glucagon secretion. Studies in diabetic rats indicate that the physiological counter-regulatory response is suppressed in insulin-treated diabetes, a defect that can be corrected by somatostatin antagonists.

The DEPTH trial will test the novel hypothesis that hypoglycaemia results from hypersecretion of somatostatin, and that this defect can be corrected by SGLT2i. As these medications are already in clinical use, our findings may be rapidly translated into practice. Understanding these key processes has the potential to generate novel therapeutic strategies to improve glycaemic control, thereby facilitating a more active lifestyle in people with T1DM.

DETAILED DESCRIPTION:
PART A Study visit 1 (30min, day 1): 1. Observations documented in CRF: resting heart rate and blood pressure 2. CGM sensor inserted. 3. Insulin dose reduced by approximately 15%. 4. Participants instructed to return on day 3 (study visit 2) fasted (no breakfast), and to refrain from exercising until then. 5. If they experience a hypoglycaemic episode within 24h of visit 2 then it will be postponed by 2 days. The medical research team will review the participant's insulin dose and make any required changes. If following this a second hypoglycaemia event occurs, then the participant will be withdrawn from the trial.

Study visit 2 (5 hours, day 3): 1. Observations documented in CRF: resting heart rate and blood pressure 2. Euglycaemic clamp for up to 1.5h to maintain blood glucose at 5mmol/L (90mg/dL) 3. Exercise challenge 4. If a participant fails to reach hypoglycaemia (defined as <3.3mmol/L, 60mg/dL) during the exercise challenge, then the study visit will be repeated after at least 2 days of washout/rest. If they again fail to reach hypoglycaemia then they will be withdrawn from the trial. 5. If the exercise challenge is completed with a hypoglycaemia episode, then the participant will proceed to Part B.

Following visit 2, participants will be allocated to a treatment group using an adaptive randomisation scheme. This will be used to balance the groups' baseline characteristics (age, sex & fitness level) in this relatively small pilot trial.

PART B Study visit 3 (30 minutes, day 8): 1. Observations documented in CRF: resting heart rate and blood pressure 2. CGM sensor inserted (if required). 3. Participants informed which arm of the study they have been randomised to, and supplied with their prescription of dapagliflozin. Participants in arm B1 will take the single dose when they attend study visit 4. Participants in arm B2 will begin taking their regular dose of dapagliflozin immediately. 4. Participants instructed to return on day 10 (study visit 4) fasted (no breakfast), and to refrain from exercising until then. 5. If they experience a hypoglycaemic episode within 24h of visit 4 then the exercise challenge will be postponed by 2 days. The medical research team will review the participant's insulin dose and make any required changes. If following this a second hypoglycaemia event occurs, then the participant will be withdrawn from the trial.

Study visit 4 (5 hours; day 10): 1. Observations documented in CRF: resting heart rate and blood pressure 2. (Arm B1): single dose of dapagliflozin taken when they arrive at the department unless they have experienced a hypoglycaemia event earlier in the morning. (Arm B2): compliance with dapagliflozin regimen and adverse events recorded in the CRF by the medical research team. 3. Euglycaemic clamp for up to 1.5h to maintain blood glucose at 5mmol/L (90mg/dL) 4. Exercise challenge 5. Participants in Arm B2 will be instructed to take one final dose of dapagliflozin the following day. All participants will be instructed to return to their pre-trial insulin dose after 48h 6. Arrangements made for end of study visit (either at CRU or home-visit).

Study visit 5 (30min; day 12-20): 1. End of study visit (either at CRU or home-visit) 2. CGM sensor removed and data downloaded. CGM system returned to CRU. 3. (Arm B1): adverse events recorded. (Arm B2): compliance with dapagliflozin regimen, adverse events recorded and any unused dapagliflozin returned (document drug accountability).

Telephone follow-up (15min; 19-27 days after study visit 5): 1. Documentation of any adverse events occurred following the discontinuation of dapagliflozin. 2. Participant informed about end of study

ELIGIBILITY:
Inclusion criteria:

1. Age 18-74
2. T1DM diagnosed at least 12 months prior to screening test
3. On insulin pump or multiple daily injections
4. HbA1c <10% (86 mmol/L)
5. Engage in some form of regular exercise
6. Have experienced at least one episode of exercise-induced hypoglycaemia
7. Adequate treatment of celiac disease if it exists.
8. Willing and able to give informed consent for participation in the trial
9. In the Investigator's opinion is able and willing to comply with all trial requirements
10. Will allow their General Practitioner to be notified of participation in the trial.

Exclusion criteria:

1. History of seizures or coma associated with hypoglycaemia in the past 2 years.
2. Active diabetic retinopathy ( including proliferative diabetic retinopathy or vitreous haemorrhage in the past 6 months).
3. Pregnant, breastfeeding, planning to become pregnant or not using adequate contraception methods (females only) during the course of the study
4. History of ischemic heart disease ( unless has had successful reperfusion), stroke/TIA, ventricular rhythm disturbances or thromboembolic disease.
5. A history of hypotension if currently on antihypertensive therapy
6. An episode of diabetic ketoacidosis in the previous 1 month
7. Currently on loop diuretics
8. On beta-blocker medication
9. A history of heart failure (NYHA Class 3 or 4)
10. A history of rare hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose-galactose malabsorption
11. Renal impairment ( eGFR<60 ml/min/1.73m2)
12. Untreated Graves disease
13. ECG or stress test findings indicating active ischemia or a condition that would compromise the participant's safety
14. Major psychiatric disease including diagnosed eating disorders, history of drug or alcohol abuse.
15. Known or suspected allergy to trial medication
16. Oral or injectable steroid treatment 30 days prior to the start or at any time during the trial period
17. Known malignancy or any other condition or circumstances which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol.
18. Receipt of any investigational trial drug within 3 months prior to participation in the current trial.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Time to hypoglycaemia during the exercise challenge, before and after dapagliflozin treatment. | 90min exercise challenge during Part A and Part B
  To determine whether dapagliflozin (either regular or as a single dose) can delay/prevent the onset of hypoglycaemia during moderate intensity exercise.
  Following blood glucose stabilisation at 5mmol/L (90mg/dL) during the euglycaemic clamp, participants will begin exercising at moderate intensity (50-60% VO2 max) for up to 90min. Time to hypoglycaemia (defined as blood glucose <3.3mmol/L, 60mg/dL) will be determined before (Part A) and after (Part B) dapagliflozin treatment.

SECONDARY OUTCOMES:
Duration of time in hypoglycaemia following the exercise challenge, before and after dapagliflozin treatment. | 24-hour period after each exercise challenge
  To determine whether dapagliflozin can prevent late-onset exercise-induced hypoglycaemia (categorised as <4mmol/L or <3mmol/L from continuous glucose monitoring recordings) overnight or the following day, before and after dapagliflozin treatment and between treatment groups (B1: single dose; B2: regular dose).
Concentration of plasma glucose, glucagon and somatostatin-14 at each 10min interval during the exercise challenge. | Every 10min during the 90min exercise challenge during Part A and Part B
  To characterise the secretion of glucagon and somatostatin during and after exercise, on and off dapagliflozin.
  The concentration of plasma glucose, glucagon and somatostatin-14 (pancreatic- specific) at each 10min interval during the exercise challenge will be measured before (Part A) and after (Part B) dapagliflozin treatment.
Concentration of plasma potassium, sodium, calcium and pH at each 10min interval during exercise challenge | Every 10min during the 90min exercise challenge during Part A and Part B
  To determine the plasma electrolyte changes during exercise.
  The concentration of plasma potassium, sodium, calcium and pH at each 10min interval during exercise challenge will be measured before (Part A) and after (Part B) dapagliflozin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Spiliotis, MD, Principal Investigator — University of Oxford
Locations (1):
- Clinical Research Unit, OCDEM, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes